CLINICAL TRIAL: NCT07146256
Title: Natural History of Oculo-Pharyngeal Muscular Dystrophy (OPMD) - Israel National OPMD Registry
Acronym: Isr-OPMD
Status: Recruiting | Type: Observational
Sponsor: Sheba Medical Center (Other Government)
Collaborators: The non-profit organization for promotion of health and cure of OPMD (Unknown)
Responsible Party: Sponsor
Other Study IDs: SHEBA-21-8801-AD-CTIL
Record Dates: First submitted 2025-08-05; First posted 2025-08-28 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Oculopharyngeal Muscular Dystrophy (OPMD)
Keywords: Oculopharyngeal muscular dystrophy (OPMD); Natural history; Dysphagia; Eyelid ptosis; Muscle weakness; Oral health
MeSH Terms: conditions — Muscular Dystrophy, Oculopharyngeal; Deglutition Disorders; Blepharoptosis; Muscle Weakness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Subjects with genetically diagnosed OPMD
  Interventions: Other: Non-interventional observational study

INTERVENTIONS:
Other: Non-interventional observational study — No intervention will be studied

SUMMARY:
The goal of this open prospective multi-disciplinary observational study of patients with OPMD at various stages of clinical manifestations is to explore the natural history of the disease in the Israeli population.

DETAILED DESCRIPTION:
The the following procedures will be performed by a multidisciplinary team:

Neurological and neurocognitive examination; Clinical assessment of of swallowing and severity of dysphagia; Clinical assessment of eyelid ptosis severity; Clinical assessment of respiratory muscles function; Clinical assessment of oral health

ELIGIBILITY:
Inclusion Criteria:

* Patients with clinical diagnosis of OPMD or patients with signs /symptoms suggestive of OPMD

Exclusion Criteria:

* Age <18 years and Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Genetically Confirmed Oculopharyngeal Muscular Dystrophy
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2030-01 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
Severity of muscle strength decline over time | 1 year
  10-meter walk test
Penetration/Aspiration Scale | 1 year
  Penetration/Aspiration Scale (PAS)
Upper Margin Reflex Distance | 1 year
  Upper Margin Reflex Distance
Lower Margin Reflex Distance | 1 year
  Lower Margin Reflex Distance

SECONDARY OUTCOMES:
Maximum Expiratory Pressure | 2 years
  Maximum Expiratory Pressure (MEP)
Cough Peak Flow | 2 years
  Cough Peak Flow (CPF)
Oral health | 2 years
  Decayed, Missing, and Filled Teeth (DMFT) index
Dysphagia severity | 1 year
  Yale Pharyngeal Residue Severity Rating Scale
Functional Oral Intake Scale | 1 year
  Functional Oral Intake Scale (FOIS)
Swallowing Disturbance | 1 year
  Swallowing Disturbance Questionnaire (SDQ)

CONTACTS AND LOCATIONS:
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel

REFERENCES:
- See also: The National Israeli Registry for Oculo-Pharyngeal Muscular Dystrophy (IsrO-PMD): rationale and design — https://doi.org/10.1007/s44162-023-00020-z